CLINICAL TRIAL: NCT02012192
Title: A Two-part, Multicentre, International Phase I and II Trial Assessing the Safety and Efficacy of the Hsp90 Inhibitor Ganetespib in Combination With Paclitaxel Weekly in Women With High-grade Serous, High-grade Endometrioid, or Undifferentiated, Platinum-resistant Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: GANNET53: Ganetespib in Metastatic, p53-mutant, Platinum-resistant Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: production of IMP has stopped
Sponsor: Medical University Innsbruck (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Nicole Concin, Univ.-Prof. Dr., Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GANNET53; 2013-003868-31 (EudraCT Number)
Record Dates: First submitted 2013-12-02; First posted 2013-12-16 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-06

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: High-grade serous; high-grade endometrioid; undifferentiated
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Disorders of Sex Development | interventions — STA 9090; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ganetespib + Paclitaxel (Experimental): Drug: ganetespib, dose will depend on phase I results, given iv once weekly for 3 out of 4 weeks (days 1, 8, 15 of each 4-weeks/28-days cycle); Drug: paclitaxel, 80 mg/m2, given iv once weekly for 3 out of 4 weeks (days 1, 8, 15 of each 4-weeks/28-days cycle), until progression.
  Interventions: Drug: Ganetespib; Drug: Paclitaxel
- Paclitaxel (Active Comparator): Drug: paclitaxel: 80 mg/m2, given iv once weekly for 3 out of 4 weeks (days 1, 8, 15 of each 4-weeks/28-days cycle), until progression
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Ganetespib
  Arms: Ganetespib + Paclitaxel
Drug: Paclitaxel

SUMMARY:
Epithelial ovarian cancer (EOC) is the most lethal gynaecological malignancy causing 41900 deaths annually in Europe. The predominance of aggressive Type II tumours, which are characterised by a high frequency of p53 mutations, and primary or acquired resistance to platinum-based chemotherapy profoundly contribute to the high mortality rate. With current standard therapy the median overall survival of metastatic platinum-resistant (Pt-R) ovarian cancer patients is only 14 month. There is a pressing need for more effective, innovative treatment strategies to particularly improve survival in this subgroup of EOC patients. This is a drug strategy targeting a central driver of tumour aggressiveness and metastatic ability, namely mutant p53, via an innovative new Hsp90 (heat shock protein 90) inhibition mechanism. The most advanced, second-generation Hsp90 inhibitor will be used, Ganetespib. The first part (Phase I) of the GANNET53 trial will test the safety of Ganetespib in a new combination with standard chemotherapy (Paclitaxel weekly) in Pt-R EOC patients. The second part (randomised Phase II) will examine the efficacy of Ganetespib in combination with standard chemotherapy versus standard chemotherapy alone in EOC patients with Pt-R tumours.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign and date a written informed consent document
* Female patients ≥18 years of age
* High-grade serous, high-grade endometrioid, or undifferentiated epithelial ovarian, fallopian tube or primary peritoneal cancer
* Patients in part II: High-grade serous, high-grade endometrioid, or undifferentiated epithelial ovarian, fallopian tube or primary peritoneal cancer confirmed by central histopathology through archival formalin-fixed paraffin embedded (FFPE) or fresh-frozen tumour samples.

  • Platinum-resistant disease:
* primary platinum-resistant disease: progression > 1 month and ≤ 6 months after completion of primary platinum-based therapy
* secondary platinum-resistant disease (including secondary platinum-refractory disease): progression ≤ 6 months after (or during) reiterative platinum-based therapy
* Patients must have disease that is measurable according to RECIST 1.1 or assessable according to the GCIG (Eastern Cooperative Oncology Group) CA-125 criteria
* ECOG performance status of 0-1
* Life expectancy of at least 3 months as assessed by the investigator

Adequate function of the bone marrow:

* Platelets ≥100 x 109/L
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Haemoglobin ≥ 8.5 g/dl. Patients may receive blood transfusion(s) to maintain haemoglobin values > 8.5 g/dl.

Adequate organ functions:

* Creatinine < 2 mg/dl (<177 µmol/L)
* Total bilirubin ≤ 1.5 x upper limit of normal
* SGOT ( serum glutamate oxaloacetate transaminase)/SGPT (serum glutamate pyruvate transaminase) (AST/ALT) ≤ 3 x upper limit of normal
* Urinanalysis or urine dipstick for proteinuria less than 2+. Patients with ≥ 2+ on dipstick should undergo 24-hour urine collection and must demonstrate < 1 g of protein/24 hours. Alternatively, proteinuria testing can be performed according to local standards
* Negative urine/serum pregnancy test in women of childbearing potential (WOCBP, see section 5). WOCBP who are sexually active, agree to use highly effective means of contraception during the study and for at least 6 months post-study treatment. Allowed are accepted and effective non-hormonal methods of contraception and sexual abstinence or vasectomised partners (>3 months previously). Vasectomy has to be confirmed by two negative semen analyses.
* Availability of archival ovarian cancer tissue for central histopathological review and p53 mutational analysis

Exclusion Criteria:

* Ovarian tumours with low malignant potential (i.e. borderline tumours)
* Primary platinum-refractory disease (progression during primary platinum-based chemotherapy)

PRIOR, CURRENT OR PLANNED TREATMENT:

* Previous treatment with > 2 chemotherapy regimens in the platinum-resistant setting (excluding targeted and endocrine therapies).
* More than 4 previous lines of chemotherapy.
* Major surgery within 2 weeks prior to first dose of ganetespib

PRIOR OR CONCOMITANT CONDITIONS OR PROCEDURES:

* Patients with a history of prior malignancies, except, disease-free time-frame of ≥ 3 years prior to randomisation.
* Patients with prior in-situ carcinomas, except:

complete removal of the tumour is given

* Known history of severe (grade 3 or 4) allergic or hypersensitivity reactions to excipients (e.g., polyethylene glycol [PEG] 300 and Polysorbate 80)
* History of intolerance or hypersensitivity to paclitaxel and/or adverse events related to paclitaxel that resulted in paclitaxel being permanently discontinued
* Peripheral neuropathy of grade > 2 per NCI CTCAE (Common Toxicity Criteria for Adverse Effects), version 4.03, within 4 weeks prior to randomisation
* Clinical symptomatic bowel obstruction at time of screening
* Left ventricular ejection fraction defined by MUGA (multigated acquisition)/ECHO below the institutional lower limit of normal
* Patients with symptomatic brain metastases
* Significant cardiac disease: New York Heart Association (NYHA) Class 3 or 4; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty or coronary artery bypass graft (CABG) within the past 6 month; or uncontrolled atrial or ventricular cardiac arrhythmias.
* History of prolonged QT syndrome, or family member with prolonged QT syndrome
* QTc (corrected QT interval) interval > 470 msec when 3 consecutive EKG values are averaged
* Ventricular tachycardia or a supraventricular tachycardia that requires treatment with a Class Ia antiarrhythmic drug (e.g., quinidine, procainamide, disopyramide) or Class III antiarrhythmic drug (e.g., sotalol, amiodarone, dofetilide). Use of other antiarrhythmic drugs is permitted
* Second- or third-degree atrioventricular (AV) block, except:

treated with a permanent pacemaker

* Complete left bundle branch block (LBBB)
* Any other condition that, in the opinion of the investigator, may compromise the safety, compliance of the patient, or would preclude the patient from successful completion of the study.
* Participation in another clinical study with experimental therapy within 28 days before start of treatment.
* Women who are pregnant or are lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-07-04 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Concin, MD, Principal Investigator — Medical University Innsbruck
Locations (10):
- Medical University Innsbruck, Department for Gynaecology and Obstetrics, Innsbruck, Austria
- Katholieke Universiteit Leuven, Dept. of Gynaecologic Oncology, Leuven, Belgium
- France (3):
  - Centre de lutte contre le cancer Francois Baclesse, Caen
  - Centre Anticancereux Léon Bérard, Lyon
  - Assistance Publique - Hôpitaux de Paris Medical Oncology Department, Paris
- Germany (5):
  - Universitätsmedizin Berlin Charité, Dept. for Gynecology, Berlin
  - University Hospital Carl Gustav Carus Dresden, Department of Gynaecology and Obstetrics, Dresden
  - Kliniken Essen Mitte, Evang. Huyssens-Stiftung / Knappschaft GmbH Department of Gynaecologic Oncology, Essen
  - Universitätsklinikum Hamburg-Eppendorf Dept. of Gynecology and Gynecologic Oncology, Hamburg
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Ganetespib + Paclitaxel: Drug: ganetespib, 150 mg/m², given iv once weekly for 3 out of 4 weeks (days 1, 8, 15 of each 4-weeks/28-days cycle); Drug: paclitaxel, 80 mg/m2, given iv once weekly for 3 out of 4 weeks (days 1, 8, 15 of each 4-weeks/28-days cycle), until progression.
  Ganetespib
  Paclitaxel
- Paclitaxel: Drug: paclitaxel: 80 mg/m2, given iv once weekly for 3 out of 4 weeks (days 1, 8, 15 of each 4-weeks/28-days cycle), until progression
  Paclitaxel
Period: Overall Study
Arm/Group | Ganetespib + Paclitaxel | Paclitaxel
Started | 90 | 43
Completed | 63 | 43
Not Completed | 27 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ganetespib + Paclitaxel: Drug: ganetespib, 150 mg/m², given iv once weekly for 3 out of 4 weeks (days 1, 8, 15 of each 4-weeks/28-days cycle); Drug: paclitaxel, 80 mg/m2, given iv once weekly for 3 out of 4 weeks (days 1, 8, 15 of each 4-weeks/28-days cycle), until progression.
- Total: Total of all reporting groups
Arm/Group | Ganetespib + Paclitaxel | Paclitaxel | Total
Number analyzed (Participants) | 90 | 43 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 25 | 82
  >=65 years | 33 | 18 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 43 | 133
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic group: White | 66 | 31 | 97
  Ethnic group: Black | 0 | 0 | 0
  Ethnic group: Asian | 1 | 0 | 1
  Ethnic group: Privacy | 23 | 12 | 35
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 1 | 2
  Belgium | 20 | 10 | 30
  France | 37 | 17 | 54
  Germany | 32 | 15 | 47

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: evaluate the efficacy of ganetespib in combination with weekly paclitaxel compared to weekly paclitaxel alone as measured by Progression-free survival (PFS). Response or progression will be evaluated in this study according to Response Evaluation Criteria In Solid Tumors Criteria version 1.1., CA-125 according to published GCIG criteria, and by the investigator on the basis of physical and/or gynaecological examinations.
Time Frame: Time until progression (median w/o new drug 4 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib + Paclitaxel | Paclitaxel
Number analyzed (Participants) | 90 | 43
months | 3.5 [3.092 to 3.882] | 5.3 [4.006 to 6.652]

ADVERSE EVENTS:
Time Frame: After informed consent has been obtained but prior to initiation of the study drug, only SAEs considered to be related to a protocol-mandated intervention were reported. After initiation of study drug, all AEs and SAEs regardless of relationship to the study drug, will be reported until safety follow-up at 28 days after the last dose of IMP or EOT or until the event has resolved to baseline grade or better.
Description: An AE is any untoward adverse change from the subject's baseline condition, i.e. any unfavourable and unintended sign including an abnormal laboratory finding, symptom or disease which is considered to be clinically relevant by the physician that occurs during the course of the study, whether or not considered related to the study drug.
  All AEs collected during the course of the trial (from the time of informed consent until EOT as described above) have been reported here.
Arm/Group | Ganetespib + Paclitaxel | Paclitaxel
All-Cause Mortality (participants affected / at risk) | 66/90 | 29/43
Serious Adverse Events (participants affected / at risk) | 34/90 | 10/43
Other Adverse Events (participants affected / at risk) | 88/90 | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganetespib + Paclitaxel (N=90) | Paclitaxel (N=43)
Anemia (Blood and lymphatic system disorders) | 1 | 0
febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hypovolemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal distention (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 1
Rectal Ulcer (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 8 | 1
Small intestinal perforation (Gastrointestinal disorders) | 2 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Subobstruction colon (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Fever (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 2 | 1
Infusion site extravasation (General disorders) | 0 | 1
Sudden death NOS (General disorders) | 1 | 0
Hemobilia (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Icterus (Hepatobiliary disorders) | 1 | 0
Sepsis (Infections and infestations) | 6 | 0
Urinary tract infection (Infections and infestations) | 5 | 1
Erysipelas (Infections and infestations) | 0 | 3
Catheter related infection (Infections and infestations) | 1 | 0
Urethral infection (Infections and infestations) | 1 | 0
Infection NOS (Infections and infestations) | 0 | 1
Rupture of renal pelvis (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyperptassemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Visual acuity reduced (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 0
Kidney insufficiency (Renal and urinary disorders) | 1 | 0
Renal disorders NEC (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Thromboemblic events (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ganetespib + Paclitaxel (N=90) | Paclitaxel (N=43)
Anemia (Blood and lymphatic system disorders) | 56 | 27
Abdominal pain (Gastrointestinal disorders) | 31 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 8 | 2
Constipation (Gastrointestinal disorders) | 21 | 9
Diarrhea (Gastrointestinal disorders) | 73 | 15
Dry mouth (Gastrointestinal disorders) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 | 2
Mucositis oral (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 41 | 21
Vomiting (Gastrointestinal disorders) | 29 | 9
Astenia (General disorders) | 22 | 11
Edema limbs (General disorders) | 7 | 4
Edema peripheral (General disorders) | 6 | 7
Fatigue (General disorders) | 26 | 8
Fever (General disorders) | 10 | 0
Malaise (General disorders) | 0 | 3
Mucosal inflammation (General disorders) | 5 | 0
Allergic reaction (Immune system disorders) | 5 | 3
Bronchial infection (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 8 | 6
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 3
Electrocardiogram QT corrected intervall prolonged (Investigations) | 13 | 0
Lymphocyte count decreased (Investigations) | 9 | 4
Neutrophil count decreased (Investigations) | 26 | 10
Weight loss (Investigations) | 9 | 0
White blood cells decreased (Investigations) | 13 | 6
Anorexia (Metabolism and nutrition disorders) | 18 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 3
Anthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 10 | 2
Neuropath peripheral (Nervous system disorders) | 35 | 21
Paresthesia (Nervous system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 16 | 4
Cystitis non-infective (Renal and urinary disorders) | 0 | 3
Common cold (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 4
Nail infection NOS (Skin and subcutaneous tissue disorders) | 0 | 2
Flushing (Vascular disorders) | 0 | 3
Hot flashes (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 5 | 0
Lymphedema (Vascular disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT02012192/Prot_SAP_000.pdf